CLINICAL TRIAL: NCT01677117
Title: Clinical Studies of the Effects of Extracorporeal Membrane Oxygenation for Severe ARDS Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Physician of Zhongda Hospital, Southeast University, China
Other Study IDs: ECMO treatment
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: ECMO Treatment

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Acute respiratory distress syndrome (acute respiratory distress syndrome, ARDS) fatality rate can be as high as 20% -41%, once progress is severe of ARDS, mortality rose to 90%, the main cause of death was refractory hypoxemia. Mechanical ventilation as the main measure to improve hypoxemia cannot correct all hypoxemia and relating complications of mechanical ventilation, mechanical ventilation in the treatment of severe ARDS has gradually been challenged. Extracorporeal membrane oxygenation（ECMO) technology matures, so that clinicians have more choices in the face of hypoxemia, and with the deepening understanding of ECMO, ECMO may become severe ARDS first-line treatment. Currently, ECMO therapy has been recognized by the majority of medical workers. Therefore, we assume that accurately grasping the ECMO indications and standardizing the implementation of treatment can significantly improve the prognosis, shorter hospital stays, lower hospitalization costs.

ELIGIBILITY:
Inclusion Criteria:

(1) age 18-70 years; (2) severe respiratory dysfunction (Murry score ≥ 3 points or clinical optimized ventilation conditions pH remains <7.2 patients); (3) PaCO2/FiO2 <100mmHg; (4) plateau pressure >30cmH2O more than 6h，duration of no more than seven days; (5) with severe respiratory dysfunction etiology reversible.

Exclusion Criteria:

(1) high levels pressure mechanical ventilation (PEEP> 15-20cmH2O and / or Pplat> 35-40cmH2O) over 7 days; (2) continued to receive high concentrations of oxygen (FiO2> 80%) is more than 7 days; (3) severe active bleeding; (4) within 24 hours of the surgery or head injury with intracranial bleeding; (5) a variety of serious irreversible state; (6) malignancy; (7) progressive pulmonary fibrosis; (8) can not surgical problems; (9) due to cardiac dysfunction leading to ARDS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe ARDS patients
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-08; Study Completion 2012-12 (Estimated)